CLINICAL TRIAL: NCT01637883
Title: Efficacy of Benzydamine Hydrochloride Dripping at Endotracheal Tube Cuff for Prevention of Postoperative Sore Throat
Brief Title: Benzydamine HCl for Postoperative Sore Throat
Acronym: POST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Associate Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 54-039-08-1-2
Record Dates: First submitted 2012-07-07; First posted 2012-07-11 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: For Intervention
Keywords: benzydamine HCl; endotracheal tube; postoperative sore throat
MeSH Terms: interventions — Benzydamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nothing (No Intervention): nothing will be dripped on the cuff of the endotracheal tube in the control group
- benzydamine HCl (Experimental): benzydamine HCl will be dripped on the cuff of the endotracheal tube 5 minutes before induction of general anesthesia
  Interventions: Drug: benzydamine HCl

INTERVENTIONS:
Drug: benzydamine HCl — 3 ml (4.5 mg) of benzydamine hydrochloride will be dripped on the cuff of the endotracheal tube 5 minutes prior to induction of general anesthesia
  Other Names: Difflam
  Arms: benzydamine HCl

SUMMARY:
To evaluate the analgesic effect of benzydamine hydrochloride dripping on the endotracheal tube cuff for postoperative sore throat.

DETAILED DESCRIPTION:
The investigators will assign patients into either the benzydamine hydrochloride or the control group. The whole ETT cuff will be either dripped with 3 ml (4.5 mg) of benzydamine hydrochloride or nothing 5 minutes prior to anesthesia induction. The incidence and severity of POST at 0, 2, 4, 6, 12 and 24 hours postoperatively will be assessed. The potential adverse effects of benzydamine hydrochloride (throat numbness, throat burning sensation, dry mouth and thirst) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* ASA status I-II
* Mallampati grade I-II
* Duration of surgery less than 4 hours
* Patients placed in the supine position

Exclusion Criteria:

* Undergoing oral, cervical spine or thyroid surgery
* More than one attempt of ETT intubation or intubated with a technique of rapid sequence induction with cricoid pressure
* Insertion of nasogastric/orogastric tube or esophageal stethoscope
* Complaint of sore throat or hoarseness
* Presence of upper respiratory tract infection within 7 days prior to the operation
* Gastroesophageal reflux
* Known allergy to benzydamine hydrochloride or other nonsteroidal anti-inflammatory drugs (NSAIDs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
analgesic effect | 24 hours
  evaluate pain score for sore throat at 0, 2, 4, 6, 12 and 24 hours after the operation

SECONDARY OUTCOMES:
side effects of benzydamine hydrochloride | 24 hours
  the incidence of throat numbness, throat burning sensation, dry mouth and thirst)within 24 hours after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Sasikaan - Nimmaanrat, MD, Principal Investigator — Faculty of Medicine, Prince of Songkla University, Hatyai, Songkhla 90110 Thailand
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand